CLINICAL TRIAL: NCT04994041
Title: Comparison of Adductor Strengthening and Pelvic Floor Muscle Strengthening Exercises on Stress Incontinence in Gym Females
Brief Title: Adductor Strengthening and Pelvic Floor Muscle Strengthening Exercises on Stress Incontinence in Gym Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0415 Irum
Record Dates: First submitted 2021-08-05; First posted 2021-08-06 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Urinary Incontinence, Stress
Keywords: Urinary Incontinence, Pelvic Floor Exercises
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor muscle plus adductor strengthening (Experimental): pelvic floor muscle plus adductor strengthening
  Interventions: Other: Pelvic floor muscle plus adductor strengthening
- Pelvic floor muscle exercises (Active Comparator): pelvic floor muscle exercises
  Interventions: Other: Pelvic floor muscle exercises

INTERVENTIONS:
Other: Pelvic floor muscle plus adductor strengthening — 20 sessions of pelvic floor muscle strengthening plus adductor is strengthening
  Arms: Pelvic floor muscle plus adductor strengthening
Other: Pelvic floor muscle exercises — 20 sessions of pelvic floor muscle strengthening
  Arms: Pelvic floor muscle exercises

SUMMARY:
Stress incontinence is common form of urinary incontinence in females. The theme is to test if pelvic floor muscle training can be augmented by incorporating adductor muscle strengthening. Group A: with pelvic floor muscle strengthening plus adductor is strengthening. Group B: with pelvic floor muscle strengthening.

DETAILED DESCRIPTION:
Stress incontinence is common form of urinary incontinence in females. When it develops in gym doing women, it badly affects their performance and result in psychosocial problems in addition to the barriers that already have been resulted from incontinence. This study combines simple regime of hip adductor a strengthening with pelvic floor muscles. The theme is to test if pelvic floor muscle training can be augmented by incorporating adductor muscle strengthening. If this comes out to be effective, this can be great contribution to gym doing females to improve their urinary incontinence related impairments. Woman would be encouraged to continue regular exercise. This will be randomized clinical trial. There are two groups for the compression of adductors strengthening and pelvic floor muscle strengthening. Group A: with pelvic floor muscle strengthening plus adductor is strengthening. Group B: with pelvic floor muscle strengthening. The collected data will be entered in Statistical Package for the Social Sciences 20.0, Descriptive and Inferential statists will be applied. Results and conclusion will be drawn.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25-45 years of age
* Engaged in gym exercises
* Fulfilling signs and symptoms of stress incontinence

Exclusion Criteria:

* Pregnant females
* Females having any history of trauma
* Any neurological disorders affecting bowl bladder
* Any malignancy in lower abdominal area

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Urinary Distress Inventory (UDI-6) | 8 weeks
  It is 6 point scale No= 0, Not at all= 1, Somewhat= 2, Moderately= 3, Quite a bit= 4.
  Add all scores and multiply by 6 then multiply by 25 for the scale score
  The UDI-6 Total Score of 33.33 was determined to be the optimal cutoff for distinguishing between symptomatic and asymptomatic women.
  For UDI-6 scores more than 33.33 indicate higher distress caused by urinary incontinence symptoms.
The Revised Urinary Incontinence Scale (RUIS) | 8 weeks
  It is a 5 point scale with each point contain 3 to 4option.
  Possible score range of 0 - 16
  A score of less than 4 indicates that the patient has no urinary incontinence
  a score of 4-8 is considered mild.
  a score of 9-12 is considered moderate.
  a score of 13 or above is considered severe.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Riphah International University
Locations (1):
- Genesis fitness centere, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schneeweiss J, Koch M, Umek W. The human urinary microbiome and how it relates to urogynecology. Int Urogynecol J. 2016 Sep;27(9):1307-12. doi: 10.1007/s00192-016-2944-5. Epub 2016 Jan 25. PMID 26811114
- [Background] Al-Mukhtar Othman J, Akervall S, Milsom I, Gyhagen M. Urinary incontinence in nulliparous women aged 25-64 years: a national survey. Am J Obstet Gynecol. 2017 Feb;216(2):149.e1-149.e11. doi: 10.1016/j.ajog.2016.09.104. Epub 2016 Oct 6. PMID 27720862
- [Background] Oliveira M, Ferreira M, Azevedo MJ, Firmino-Machado J, Santos PC. Pelvic floor muscle training protocol for stress urinary incontinence in women: A systematic review. Rev Assoc Med Bras (1992). 2017 Jul;63(7):642-650. doi: 10.1590/1806-9282.63.07.642. PMID 28977091
- [Background] Pizzoferrato AC, Fauconnier A, Fritel X, Bader G, Dompeyre P. Urethral Closure Pressure at Stress: A Predictive Measure for the Diagnosis and Severity of Urinary Incontinence in Women. Int Neurourol J. 2017 Jun;21(2):121-127. doi: 10.5213/inj.1732686.343. Epub 2017 Jun 21. PMID 28673060
- [Background] de Mattos Lourenco TR, Matsuoka PK, Baracat EC, Haddad JM. Urinary incontinence in female athletes: a systematic review. Int Urogynecol J. 2018 Dec;29(12):1757-1763. doi: 10.1007/s00192-018-3629-z. Epub 2018 Mar 19. PMID 29552736
- [Background] Diokno AC, Newman DK, Low LK, Griebling TL, Maddens ME, Goode PS, Raghunathan TE, Subak LL, Sampselle CM, Boura JA, Robinson AE, McIntyre D, Burgio KL. Effect of Group-Administered Behavioral Treatment on Urinary Incontinence in Older Women: A Randomized Clinical Trial. JAMA Intern Med. 2018 Oct 1;178(10):1333-1341. doi: 10.1001/jamainternmed.2018.3766. PMID 30193294
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322